CLINICAL TRIAL: NCT00364234
Title: Low Magnitute Mechanical Stimuli Effects on Bone Structure in ESRD
Brief Title: Low Magnitude Mechanical Stimuli Effects on Bone Structure in ESRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Mary Leonard, MD, MSCE, Associate Professor of Pediatrics and Epidemiology, Children's Hospital of Philadelphia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21 DK74105 (completed); R21DK074105 (NIH)
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Renal Osteodystrophy
Keywords: Renal Osteodystrophy
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Low magnitude mechanical stimuli — 20 minutes standing on low magnitude high frequency vibrating platform

SUMMARY:
The proposed 6 month pilot and feasibility randomized trial will evaluate LMMS as an anabolic stimulus to bone in 30 adults on maintenance hemodialysis. The intervention will consist of 20 minute daily sessions in the home standing on an active LMMS platform or a placebo device that emits an audible hum suggestive of an active device. Each device contains an electronic monitor that documents adherence. The study will examine trabecular bone volume fraction (bone volume/total volume, BV/TV %) and architecture using microMRI, and cortical volumetric BMD and dimensions using QCT at baseline and 6 months. The hypothesis is that active LMMS will results in greater mean changes in trabecular and cortical parameters in hemodialysis patients. The proposed study will test the feasibility of conducting the intervention in dialysis patients and will generate preliminary data on rates of change in trabecular and cortical parameters in the active and placebo groups.

DETAILED DESCRIPTION:
Renal osteodystrophy (ROD) is a multifactorial and pervasive disorder in chronic kidney disease (CKD). As renal failure progresses, ensuing abnormal parathyroid hormone (PTH) secretion and mineral metabolism result in sclerosis of trabecular bone, thinning of cortical bone, and increased cortical porosity.(1) Despite the widespread use of phosphate binders and vitamin D therapies, hip fracture rates and mortality risk following fractures are markedly greater in dialysis patients, compared with the general population.

The vast majority of studies of bone loss in CKD relied on dual energy x-ray absorptiometry (DXA) measures of bone mineral density (BMD). However, DXA summarizes the total bone mass within the projected bone area, concealing disease effects on trabecular and cortical bone. For example, in high-turnover ROD, increased trabecular volume may offset cortical bone loss, resulting in normal or increased areal-BMD despite poor bone strength. Quantitative computed tomography (QCT) enables discrete assessment of trabecular and cortical volumetric BMD and dimensions. However, this is an incomplete solution in the setting of CKD because QCT does not assess trabecular architecture. Micro-magnetic resonance imaging (µMRI) provides a non-invasive technique to assess trabecular architecture. The µMRI data are quantified by 3D digital processing methods, such as topological analysis, to determine trabecular properties. Our pilot study of µMRI in dialysis patients revealed significant reductions in cortical thickness and suggested deterioration in the trabecular network. This innovative imaging modality may be uniquely suited to the assessment of ROD therapies.

Mechanical forces on the skeleton arise from muscle contraction and these forces generate signals that modulate bone architecture. Animal studies demonstrated that daily exposure to low magnitude mechanical stimuli (LMMS) enhanced trabecular and cortical bone quantity and quality. A randomized trial of LMMS in post-menopausal women demonstrated that LMMS were associated with increased DXA BMD, without adverse effects. LMMS may be uniquely suited to restore cortical and trabecular bone structure in ROD.

The study will enroll adults, ages 21-65 years, treated with maintenance hemodialysis at UPENN. The study will exclude the elderly and subjects with major co-morbid conditions in order to increase the likelihood that subjects will complete the 6 month intervention without significant interruptions due to hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* ages 21-65 years
* Maintenance Hemodialysis

Exclusion Criteria:

* Active Malignancy
* History of myocardial infarction
* Congestive heart failure III-IV stage
* Cerebrovascular disease
* Planned relocation
* Pregnancy
* Anticipated living-donor transplantation within the coming 6 months
* Liver failure
* Neuropathies
* Prior lower extremity amputation or difficult with ambulation
* History of hip fracture
* History of hip replacement
* History of orthostatic hypotension or a balance disorder
* History of a fall within 6 months prior to enrollment
* Difficulty in ambulation will be defined as difficulty climbing two flights of stairs or walking three blocks
* Patients with pacemaker or other metal implants that are contraindicated for MRI scans
* Weight > 113kg
* HIV Positive

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-05; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Trabecular Microarchitecture | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary B Leonard, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia , Philadelphia, Pennsylvania, United States
Locations (1):
- Childen's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States